CLINICAL TRIAL: NCT01070056
Title: Practice-based Trial of Blood Pressure Control in African Americans
Acronym: TLC-Clinic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Columbia University (Other); Hebrew Home at Riverdale (Other); New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HL087301-01 (NIH)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension; Physical Activity; Diet; Medication Adherence
Keywords: Blood Pressure; Lifestyle Changes; African American
MeSH Terms: conditions — Hypertension; Motor Activity; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Patients randomized to the Usual Care (UC) condition will receive standard hypertension (HTN) treatment recommendations as determined by their physicians. In addition, they will receive a 30-minute individual counseling session on therapeutic lifestyle modification, similar to PREMIER. We feel obligated ethically to provide this minimal intervention to patients in the UC group given that counseling on TLC is a standard recommendation for treatment of hypertension. To match the MINT-TLC group for content of intervention material, those in the UC group will receive print versions of the intervention materials.
  Interventions: Behavioral: Usual Care
- Therapeutic Lifestyle Changes (MINT-TLC) (Experimental): This intervention is based on established clinical practice guidelines for prevention and treatment of hypertension (HTN), which recommends weight loss (if overweight), limiting sodium and alcohol intake, regular physical activity, reducing alcohol intake, and eating a low-fat diet that is rich in fruit and vegetables. MINT-TLC will be conducted by trained research personnel. Patients will attend 10 classes over 12 weeks (intensive phase) followed by individual monthly MINT sessions for 3 months (maintenance phase). We chose the intervention schedules to pattern after the methodology of therapeutic lifestyle interventions with proven efficacy in hypertensive patients, specifically, Trial of Nonpharmacologic Approaches in Elderly Hypertensives (TONE) and PREMIER trials.
  Interventions: Behavioral: Therapeutic Lifestyle Changes (MINT-TLC)

INTERVENTIONS:
Behavioral: Therapeutic Lifestyle Changes (MINT-TLC) — This intervention is based on established clinical practice guidelines for prevention and treatment of hypertension(HTN), which recommends weight loss (if overweight), limiting sodium and alcohol intake, regular physical activity, reducing alcohol intake, and eating a low-fat diet that is rich in fruit and vegetables. MINT-TLC will be conducted by trained research personnel. Patients will attend 10 classes over 12 weeks (intensive phase) followed by individual monthly MINT sessions for 3 months (maintenance phase). We chose the intervention schedules to pattern after the methodology of therapeutic lifestyle interventions with proven efficacy in hypertensive patients, specifically, Trial of Nonpharmacologic Approaches in Elderly Hypertensives (TONE) and PREMIER trials.
  Arms: Therapeutic Lifestyle Changes (MINT-TLC)
Behavioral: Usual Care — Patients randomized to the Usual Care (UC) condition will receive standard hypertension (HTN) treatment recommendations as determined by their physicians. In addition, they will receive a 30-minute individual counseling session on therapeutic lifestyle modification, similar to PREMIER. We feel obligated ethically to provide this minimal intervention to patients in the UC group given that counseling on TLC is a standard recommendation for treatment of hypertension. To match the MINT-TLC group for content of intervention material, those in the UC group will receive print versions of the intervention materials.
  Arms: Usual Care

SUMMARY:
Poorly controlled hypertension (HTN) remains one of the most significant public health problems in the United States, in terms of morbidity, mortality, and economic burden. Despite compelling evidence supporting the beneficial effects of therapeutic lifestyle changes (TLC) on blood pressure (BP) reduction, their effectiveness remains untested in primary care practices, especially among minority patients who share a greater burden of HTN-related outcomes including chronic kidney disease, stroke and heart failure. This randomized controlled trial offers a unique opportunity to address this gap in the literature. Among 200 hypertensive African-Americans who receive care in community- based primary care practices, we will test the effectiveness of a culturally-tailored comprehensive therapeutic lifestyle intervention, delivered through group-based counseling and motivational interviewing (MINT-TLC) vs. Usual Care (UC). MINT-TLC is designed to help patients make appropriate TLC and develop skills to maintain these changes long-term. Patients in the MINT-TLC group will attend weekly group classes focused on TLC for 12 weeks (intensive phase); followed by individual motivational interviewing (MINT) sessions for 3 months (maintenance phase). Trained research personnel will deliver MINT-TLC with appropriate treatment fidelity procedures. Patients in the UC condition will receive a single individual counseling session on TLC and print versions of the intervention materials. The primary outcome is within-patient change in both systolic and diastolic blood pressure from baseline to 6 months. Secondary outcomes are levels of targeted therapeutic lifestyle behaviors; and proportion of patients with adequate blood pressure control at 6 months

DETAILED DESCRIPTION:
We will test the effectiveness of a primary care practice-based comprehensive therapeutic lifestyle intervention, delivered through group-based counseling and motivational interviewing (MINT-TLC) in a two-arm, randomized controlled trial (RCT) in 200 low-income, poorly controlled hypertensive African-American patients. MINT is a directive, participant-centered, counseling approach for initiating and maintaining behavior change that has proven effective in improving adherence to various health behaviors. We hypothesize that among African Americans with poorly controlled hypertension (HTN), those randomized to TLC group, compared to those randomized to UC, will exhibit a greater reduction in systolic and diastolic blood pressure (BP); greater levels of physical activity; percent change in weight; increased intake of fruits and vegetables; and reduced 24-hour urinary sodium excretion at 6 months.The primary outcome is within-patient change in systolic (SBP) and diastolic (DBP) from baseline to 6 months. The secondary outcomes are the levels of physical activity, percent change in weight, dietary intake of fruits and vegetables, 24-hour urinary sodium excretion and BP control rates at 6 months. Blood pressure will be assessed with a well-validated automated digital BP monitor (BPTru), following American Heart Association guidelines. Therapeutic lifestyle behaviors will be assessed with validated self-report measures: Dietary intake will be assessed with the NCI's fruit/vegetable and fat brief dietary assessment questionnaires; and physical activity will be assessed with the Nurses Health Study and Health Professionals Study's physical activity questionnaire. Percent weight loss will be estimated from the difference in weight between baseline and 6 months, while 24-hour urinary sodium excretion will be used to estimate dietary sodium intake. Patients are categorized as having controlled BP if their average BP that fulfills the Seventh Joint National Committee on Detection, Evaluation and Treatment of Hypertension (JNC-7) criteria of SBP < 130 and DBP < 80 mmHg (patients with diabetes or chronic kidney disease); or SBP < 140 and DBP < 90 mmHg (for all other patients). Regardless of group assignments, all outcomes data will be assessed at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Receiving care within the NYU Ambulatory Care Network for at least one year.
* Patient must have uncontrolled HTN defined as an average SBP≥140 mmHg or DBP≥90 mmHg (SBP≥130 mmHg or DBP≥80 mmHg for patients with diabetes or chronic kidney disease) on at least two previous visits in the past year
* English speaking
* Self-identify as Black, or African American;
* Permission by patient's physician to participate in the study.
* CARE-DIAG score < 6 (participants age 60 and older only)

Exclusion Criteria:

* Being deemed unable to comply with the study protocol (either self-selected or by indicating during screening that s/he could not complete all requested tasks including attend intervention classes if he/she were to be randomized to the intervention group).
* Participation in other clinical trials.
* Diagnosis of cognitive dysfunction or significant psychiatric comorbidity (as indicated in medical record).
* Blood pressure reading ≥ 180/110 at initial screening/baseline visit
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is within-patient change in systolic (SBP) and diastolic (DBP) from baseline to 6 months. | 6 months

SECONDARY OUTCOMES:
The secondary outcomes are the levels of physical activity, percent change in weight, dietary intake of fruits and vegetables, 24-hour urinary sodium excretion and BP control rates at 6 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gbenga G Ogedegbe, M.D., Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - Woodhull Medical & Mental Health Center, Brooklyn, New York
  - Governeur Hospital, New York, New York
  - Bellevue Hospital Center, New York, New York
  - Lincoln Hospital and Harlem Hospital, New York, New York

REFERENCES:
- [Derived] Ogunlade AO, Williams SK, Joseph J, Onakomaiya DO, Eimicke JP, Teresi JA, Williams O, Ogedegbe G, Spruill TM. Prevalence and correlates of depression among black and Latino stroke survivors with uncontrolled hypertension: a cross-sectional study. BMJ Open. 2020 Dec 8;10(12):e040461. doi: 10.1136/bmjopen-2020-040461. PMID 33293392
- [Derived] Schoenthaler A, Luerassi L, Silver S, Odedosu T, Kong J, Ravenell J, Teresi JA, Ogedegbe G. Comparative Effectiveness of a Practice-Based Comprehensive Lifestyle Intervention vs. Single Session Counseling in Hypertensive Blacks. Am J Hypertens. 2016 Feb;29(2):280-7. doi: 10.1093/ajh/hpv100. Epub 2015 Jul 1. PMID 26135553
- [Derived] Schoenthaler A, Luerassi L, Teresi JA, Silver S, Kong J, Odedosu T, Trilling S, Errico A, Uvwo O, Sebek K, Adekoya A, Ogedegbe G. A practice-based trial of blood pressure control in African Americans (TLC-Clinic): study protocol for a randomized controlled trial. Trials. 2011 Dec 22;12:265. doi: 10.1186/1745-6215-12-265. PMID 22192273